CLINICAL TRIAL: NCT00241605
Title: AVANDAMET Compared to Metformin Evaluation Trial (ACME): A 48-week Randomized, Open-label, Multicenter Study to Compare the Efficacy and Tolerability of AVANDAMET to Metformin Monotherapy in Subjects With Type 2 Diabetes Mellitus Who Are Not Achieving Glycemic Control on Submaximal Metformin.
Brief Title: AVANDAMET Versus Metformin For Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 712753/008
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metformin; AVANDAMET; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — rosiglitazone-metformin combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosiglitazone/metformin

SUMMARY:
This 48-week study will compare AVANDAMET vs. Metformin monotherapy for blood glucose control in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years of age with Type 2 Diabetes Mellitus and are currently on metformin monotherapy for glycemic control (100mg daily for at least 3 months prior to screening).
* Patients must have stopped previous treatment with thiazolidinediones or other anti-diabetic agents at least 3 months prior to screening.
* Women must be post-menopausal, surgically sterile or using acceptable contraceptive measures.

Exclusion Criteria:

* Prior history of hepatocellular reaction to or severe edema associated with the use of thiazolidinediones.
* Have a known hypersensitivity to thiazolidinediones or biguanides.
* Currently using insulin or any oral anti-diabetic agent other than metformin.
* History of metabolic acidosis.
* History of substance abuse.
* Have active cancer other than localized squamous or basal cell carcinoma.
* Chronic disease requiring treatment with corticosteroids.
* Other criteria will be evaluated at the screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-06-25; Primary Completion 2005-12-01 (Actual); Study Completion 2005-12-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at week 48.

SECONDARY OUTCOMES:
Change from baseline in FPG at week 48. Time to glycemic control. Change from baseline in C-peptide and insulin at week 48.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (67):
- Canada (67):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Medicine Hat, Alberta
  - GSK Investigational Site, Aldergrove, British Columbia
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Fredericton, New Brunswick
  - GSK Investigational Site, Houston, New Brunswick
  - GSK Investigational Site, Neguac, New Brunswick
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Carbonear, Newfoundland and Labrador
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Dartmouth, Nova Scotia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Upper Tantallon, Nova Scotia
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Cambridge, Ontario
  - GSK Investigational Site, Fort Erie, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Innisfil, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, North York, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Rexdale, Ontario
  - GSK Investigational Site, Richmond Hill, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Smiths Falls, Ontario
  - GSK Investigational Site, Sutton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Woodbridge, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Brossard, Quebec
  - GSK Investigational Site, Charlesbourg, Quebec
  - GSK Investigational Site, Châteauguay, Quebec
  - GSK Investigational Site, Courcelette, Quebec
  - GSK Investigational Site, Cowansville, Quebec
  - GSK Investigational Site, Hull, Quebec
  - GSK Investigational Site, Lambton, Quebec
  - GSK Investigational Site, Lle Perrot, Quebec
  - GSK Investigational Site, Longueuil, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pierrefonds, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Richelieu, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Saint-Jean-sur-Richelieu, Quebec
  - GSK Investigational Site, Saint-Léonard, Quebec
  - GSK Investigational Site, Sainte-Anne-de-Bellevue, Quebec
  - GSK Investigational Site, Sainte-Catherine, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sainte-Henri de Levis, Quebec
  - GSK Investigational Site, Salaberry-de-Valleyfield, Quebec
  - GSK Investigational Site, Thetford-Mines, Quebec
  - GSK Investigational Site, Vaudreuil, Quebec
  - GSK Investigational Site, Ville Lasalle, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
  - GSK Investigational Site, Québec